CLINICAL TRIAL: NCT06053788
Title: PocDoc Lipids Usability Study for Self-test Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vital Signs Solutions Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 322100
Record Dates: First submitted 2023-09-06; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PocDoc (Experimental): All participants given PocDoc device
  Interventions: Diagnostic Test: PocDoc

INTERVENTIONS:
Diagnostic Test: PocDoc — Point of care digital lipid test

SUMMARY:
This study seeks to expand the approved indication of use for a UKCA approved IVD device. PocDoc lipids is approved for professional use to measure the levels of lipids in a fingerprick blood samples. This study will investigate the usability of the device by untrained lay people in order to expand the device's utility to the self-test setting.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Subjects are legally competent and capable to understand character, meaning and consequences of the study
* Subjects own an approved mobile device (these will be available at the time of the study on the PocDoc website and a link will be contained in the PIS)

Exclusion Criteria:

* Being unable to give informed consent
* < 18 years or > 85 years
* Legally incompetent
* Language barriers potentially compromising an adequate compliance with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Usability | Day 1 - one single test done at one timepoint
  The usability study will pass our acceptance criteria if 95% of the users are able to successfully conduct a PocDoc lipid test, obtaining a result. The PocDoc lipid test is a rapid 5-marker lipid test in lateral flow format that uses a smartphone application to analyse and display the result.
  Usability is defined as the ability of an individual to navigate the mobile application steps to conduct the rapid lateral flow test, to take a picture of the image and to navigate to the results page of the application to see their results. A successful test is one where the individual successfully completes all steps and gets their result.

CONTACTS AND LOCATIONS:
Locations (1):
- Vital Signs Solutions Ltd, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No